CLINICAL TRIAL: NCT04687163
Title: Sorafenib or Lenvatinib Plus Hepatic Artery Infusion of 130 mg/m² Oxaliplatin, Leucovorin, and Fluorouracil Versus Sorafenib or Lenvatinib Plus Hepatic Artery Infusion of 85 mg/m² Oxaliplatin, Leucovorin, and 1200 mg/m² Fluorouracil for Unresectable Advanced Hepatocellular Carcinoma: a Randomised Phase 3 Trial
Brief Title: Sorafenib or Lenvatinib Plus HAIC of 130 mg/m² Oxaliplatin, and 5-fu vs Sorafenib or Lenvatinib Plus HAIC of 85mg/m² Oxaliplatin, and 5-fu for Unresectable Advanced HCC: a Randomised Phase 3 Trial
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Kaiping Central Hospital (Other); Guangzhou No.12 People's Hospital (Other Government)
Responsible Party: Principal Investigator, Shi Ming, Proffessor, Sun Yat-sen University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SH-3
Record Dates: First submitted 2020-12-24; First posted 2020-12-29 (Actual); Last update posted 2021-01-13 (Actual); Status verified 2020-12

CONDITIONS: Hepatocellular Carcinoma
MeSH Terms: conditions — Carcinoma, Hepatocellular | interventions — Fluorouracil

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OXA 130 (Experimental): Patients received sorafenib or lenvatinib Plus HAIC of 130 mg/m² oxaliplatin, and 2400 mg/m² 5-fu
  Interventions: Drug: HAIC of 130 mg/m² Oxaliplatin, and 5-fu; Drug: TKI
- OXA 85 (Active Comparator): Patients received sorafenib or lenvatinib Plus HAIC of 85 mg/m² oxaliplatin, and 2400 mg/m² 5-fu
  Interventions: Drug: HAIC of 85 mg/m² Oxaliplatin, and 5-fu; Drug: TKI

INTERVENTIONS:
Drug: HAIC of 130 mg/m² Oxaliplatin, and 5-fu — Hepatic arterial infusion of 130 mg/m² oxaliplatin,leucovorin and 2400 mg/m² 5-FU
  Arms: OXA 130
Drug: HAIC of 85 mg/m² Oxaliplatin, and 5-fu — Hepatic arterial infusion of 85 mg/m² oxaliplatin,leucovorin and 2400 mg/m² 5-FU
  Arms: OXA 85
Drug: TKI — sorafenib 400mg bid or lenvatinib 12 mg/day (for bodyweight ≥60 kg) or 8 mg/day (for bodyweight <60 kg)

SUMMARY:
A randomized trial showed that sorafenib plus hepatic artery infusion of 85mg/m² oxaliplatin, leucovorin and fluorouracil is more effective than sorafenib in advanced hepatocellular carcinoma. However, a retrospective study showed that hepatic artery infusion of 130 mg/m² oxaliplatin, leucovorin and fluorouracil is more effective than sorafenib in advanced hepatocellular carcinoma. It is unknown which oxaliplatin dose is better.

ELIGIBILITY:
Inclusion Criteria:

* KPS≥70;
* The diagnosis of HCC was based on the diagnostic criteria for HCC used by the European Association for the Study of the Liver (EASL).
* Patients must have at least one tumor lesion that can be accurately measured;
* With vascular invasion or extrahepatic metastasis
* Diagnosed as unresectable with consensus by the panel of liver surgery experts;
* No past history of TACE, HAIC, chemotherapy or molecule-targeted treatment;
* No Cirrhosis or cirrhotic status of Child-Pugh class A only
* Meet the following laboratory parameters:(a) Platelet count ≥ 75,000/μL; (b)Hemoglobin ≥ 8.5 g/dL;(c) Total bilirubin ≤ 30mmol/L;(d) Serum albumin

  ≥ 32 g/L;(e) ASL and AST ≤ 6 x upper limit of normal;(f) Serum creatinine

  ≤ 1.5 x upper limit of normal;(g) INR > 2.3 or PT/APTT within normal limits; (h) Absolute neutrophil count (ANC) >1,500/mm3;
* Ability to understand the protocol and to agree to and sign a written informed consent document.

Exclusion Criteria:

* Patients with clinically significant gastrointestinal bleeding within 30 days prior to study entry.
* Known of serious heart disease which can nor endure the treatment such as cardiac ventricular arrhythmias requiring anti-arrhythmic therapy
* Evidence of hepatic decompensation including ascites, gastrointestinal bleeding or hepatic encephalopathy
* Known history of HIV
* History of organ allograft
* Known or suspected allergy to the investigational agents or any agent given in association with this trial.
* Evidence of bleeding diathesis.
* Any other hemorrhage/bleeding event > CTCAE Grade 3 within 4 weeks of first dose of study drug

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 400 (Estimated)
Dates: Start 2020-12-30 (Actual); Primary Completion 2022-12-01 (Estimated); Study Completion 2022-12-01 (Estimated)

PRIMARY OUTCOMES:
Overall survival | 24 months

SECONDARY OUTCOMES:
progression-free survival | 24 months
objective response rate | 6 months
time to response | 12 months
  time to the date that patients achieved objective response
Adverse Events | 30 Days after HAIC

CONTACTS AND LOCATIONS:
Locations (3):
- China (3):
  - Cancer Center Sun Yat-sen University, Guangzhou, Guangdong
  - Guangzhou Twelfth People 's Hospita, Guangzhou, Guangdong
  - Kaiping Central Hospital, Kaiping, Guangdong